CLINICAL TRIAL: NCT04341051
Title: Sciatic Block Increases Regional Saturation in Peripheral Artery Occlusive Disease Monitored by NIRS: a Prospective Monocentric Study.
Brief Title: Sciatic Block Increases Regional Saturation in Peripheral Artery Occlusive Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Fabio Gobbi, Doctor, A.O.U. Città della Salute e della Scienza
Other Study IDs: 0033871
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Artery Occlusive Disease; Popliteal Sciatic Nerve Block
Keywords: regional oxigen saturation
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: we will observe the regional saturation of O2 through NIRS at the following time: T0(before peripheral anesthesia); T1 (5 minutes from the block); T2 (15 minutes from the block); T3 (30 minutes from the block); T4 (after revascularization); At each interval PA, SpO2 and NIRS were also recorded in the contralateral limb as control data.
  Interventions: Other: Case

INTERVENTIONS:
Other: Case — Mesure with NIRS regional saturation in patients undergoing popliteal block during vascular surgery for chronic obliterating arteriopathy (IIa to III Fontaine Classification)

SUMMARY:
We conducted Single-center prospective observational study to evaluate the improvement of peripheral vascular perfusion monitored with near-infrared spectroscopy, in patients undergoing endovascular surgery after performing sciatic nervous block.

DETAILED DESCRIPTION:
The aims of that study is to check regional oxigen saturation variability in patients suffering from Peripheral Artery Occlusive Disease (IIa to III Fontaine classification) undergoing popliteal sciatic nerve block as analgesic procedure before vascular surgery. We want to evaluate the increase in regional microcirculation after the popliteal nerve blocks due to vasoplegic response and vasodilatation after performing regional anaesthesia. We will place NIRS electrode on the instep of the foot to evaluate regional oxigen saturation in the interested leg before the performing of popliteal sciatic nerve block and then during the surgery (after 5 minuts, 15 minuts, 30 minuts), and after the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* age: > 18 years
* Peripheral artery occlusive desease involving popliteal, tibial and/or peroneal artery
* Stadiation IIa to III in Fontaine classification
* Eligibility for PTA or Stenting

Exclusion Criteria:

* trophic alteration of the application site of the NIRS
* less than 18 years
* Pregnancy
* need of sedation during the procedure
* revascularization performed as emergency surgery
* Allergic reactions with local anaesthetic
* Previous surgery involving the interested artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Peripheral Artery Occlusive Disease undergoing popliteal sciatic nerve block as analgesic procedure before revascularization surgery
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Regional Oxigen saturation downstream of popliteal region | 1 day
  NIRS misuration of delivered oxigen T0)before the execution of sciatic popliteal block T1) after 5 minuts, T2)15 minuts, T3)30 minuts, T4)after the revascularization

SECONDARY OUTCOMES:
Comparing the results between AOCP IIa to III (Fontaine Classification) | 1 day
  NIRS misuration of delivered oxigen T0)before the execution of sciatic popliteal block T1) after 5 minuts, T2)15 minuts, T3)30 minuts, T4)after the revascularization
Comparing the results between patients with occlusion of a single arthery and patients with more occluded arthery | 1 day
  NIRS misuration of delivered oxigen T0)before the execution of sciatic popliteal block T1) after 5 minuts, T2)15 minuts, T3)30 minuts, T4)after the revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Gobbi, Doctor, Principal Investigator — A.O.U. Città della Salute e della Scienza

IPD SHARING:
Plan to Share IPD: Undecided